CLINICAL TRIAL: NCT03332238
Title: A Phase II Study to Evaluate Autologous Stromal Vascular Fraction Cell Therapy to Improve the Repair of Chronically Rotator Cuff Tears
Brief Title: Stromal Vascular Fraction Cell Therapy to Improve the Repair of Rotator Cuff Tears
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-0999
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Tear; Muscle Atrophy; Tendon Tear
MeSH Terms: conditions — Rotator Cuff Injuries; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive an injection of vehicle (Ringer's solution) into their supraspinatus muscle and tendon at the time of rotator cuff repair
  Interventions: Device: Ringer's solution
- Cell Therapy (Active Comparator): Patients will receive an injection of stromal vascular fraction material suspended in vehicle (Ringer's solution) into their supraspinatus muscle and tendon at the time of rotator cuff repair
  Interventions: Device: Autologous Stomal Vascular Fraction Material

INTERVENTIONS:
Device: Autologous Stomal Vascular Fraction Material — Autologous Stomal Vascular Fraction Material Prepared from the Tissue Genesis® Icellator Cell Isolation System™
  Arms: Cell Therapy
Device: Ringer's solution — Ringer's solution
  Arms: Placebo

SUMMARY:
Rotator cuff disease is one of the most prevalent musculoskeletal conditions across the world. Patients with chronic rotator cuff tears often have substantial muscle atrophy and fatty infiltration. Surgical repair of the tear does not reverse the atrophy, and many patients continue to experience weakness, pain, and a persistent reduction in the quality of life. An important limitation in our ability to successfully rehabilitate these injuries postoperatively and return patients to normal function has to do with the poor quality of the muscle and tendon after rotator cuff repair. The stromal vascular fraction (SVF) of subcutaneous adipose tissue is highly enriched with cells (SVFCs) that can both directly participate in tissue regeneration by differentiating into myogenic and tenogenic cells, and indirectly by secreting growth factors and small molecules which activate pathways associated with healthy tissue regeneration. High numbers of autologous SVFCs can be isolated using the cost-effective, intraoperative Icellator (Tissue Genesis, Honolulu, HI) point-of-care system. This clinical trial will be determine if the use of SVFCs can enhance outcomes for patients who are undergoing surgical repair of a torn supraspinatus rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 45-65 years old at the time of enrollment
* Full-thickness supraspinatus tendon tear with endon retraction ≤ 3 cm
* Magnetic resonance imaging Goutallier score ≤ grade 2
* Completed at least 6 weeks of standard physical therapy but continue to have pain and limited function (failed physical therapy)
* Sufficient subcutaneous abdominal adipose tissue to allow the recovery of 60-120cc of lipoaspirate
* Must pass standard of care blood work screening

Exclusion Criteria:

* Any tears of any cuff tendon other than the supraspinatus
* Magnetic resonance imaging Goutallier scores ≥ 3
* Frank signs of glenohumeral osteoarthritis on magnetic resonance imaging
* A history of previous rotator cuff repair
* A history of upper extremity fracture or other moderate to severe upper extremity trauma
* A BMI < 20 or > 35
* Pregnant or breast feeding
* Premenopausal women who are not using contraception
* Previous abdominal liposuction or any major open abdominal surgery
* Type I or type II diabetes, or glycated hemoglobin (hemoglobin A1C) values > 6.5 or other metabolic disorders
* Hypercholesterolemia (total cholesterol ≥240mg/dL)
* History of cancer
* Autoimmune disorder or HIV+ status
* Use of nicotine products
* Have any other history of major medical illness, disease or other relevant orthopaedic disability
* Who do not speak English
* Liodcaine allergy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-07-23 (Estimated)

PRIMARY OUTCOMES:
Change in scapular plane abduction strength from baseline, and additional isometric, isokinetic strength measurements to assess supraspinatus function. | 2 weeks prior to surgery, 6 months after surgery, 12 months after surgery, 24 months after surgery

SECONDARY OUTCOMES:
Change in Penn Shoulder score, ASES score and Short Form Global Health scale (PROMIS-SF) from baseline (range 0 minimum to 30 maximum) | 2 weeks prior to surgery, 6 weeks after surgery, 6 months after surgery, 12 months after surgery, 24 months after surgery
Change in supraspinatus muscle stiffness from baseline, measured by ultrasound shear wave elastrography | 1 month prior to surgery, 6 months after surgery, 24 months after surgery
Change in fatty infiltration from baseline, measured by magnetic resonance imaging | 1 month prior to surgery, 6 months after surgery, 24 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rodeo, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Bedi A, Dines J, Warren RF, Dines DM. Massive tears of the rotator cuff. J Bone Joint Surg Am. 2010 Aug 4;92(9):1894-908. doi: 10.2106/JBJS.I.01531. PMID 20686065
- [Background] Mendias CL, Roche SM, Harning JA, Davis ME, Lynch EB, Sibilsky Enselman ER, Jacobson JA, Claflin DR, Calve S, Bedi A. Reduced muscle fiber force production and disrupted myofibril architecture in patients with chronic rotator cuff tears. J Shoulder Elbow Surg. 2015 Jan;24(1):111-9. doi: 10.1016/j.jse.2014.06.037. Epub 2014 Sep 3. PMID 25193488
- [Background] Davis ME, Stafford PL, Jergenson MJ, Bedi A, Mendias CL. Muscle fibers are injured at the time of acute and chronic rotator cuff repair. Clin Orthop Relat Res. 2015 Jan;473(1):226-32. doi: 10.1007/s11999-014-3860-y. Epub 2014 Aug 12. PMID 25113269
- [Background] Gumucio JP, Flood MD, Roche SM, Sugg KB, Momoh AO, Kosnik PE, Bedi A, Mendias CL. Stromal vascular stem cell treatment decreases muscle fibrosis following chronic rotator cuff tear. Int Orthop. 2016 Apr;40(4):759-64. doi: 10.1007/s00264-015-2937-x. Epub 2015 Jul 30. PMID 26224616
- [Background] Gumucio JP, Davis ME, Bradley JR, Stafford PL, Schiffman CJ, Lynch EB, Claflin DR, Bedi A, Mendias CL. Rotator cuff tear reduces muscle fiber specific force production and induces macrophage accumulation and autophagy. J Orthop Res. 2012 Dec;30(12):1963-70. doi: 10.1002/jor.22168. Epub 2012 Jun 13. PMID 22696414
- [Background] Bourin P, Bunnell BA, Casteilla L, Dominici M, Katz AJ, March KL, Redl H, Rubin JP, Yoshimura K, Gimble JM. Stromal cells from the adipose tissue-derived stromal vascular fraction and culture expanded adipose tissue-derived stromal/stem cells: a joint statement of the International Federation for Adipose Therapeutics and Science (IFATS) and the International Society for Cellular Therapy (ISCT). Cytotherapy. 2013 Jun;15(6):641-8. doi: 10.1016/j.jcyt.2013.02.006. Epub 2013 Apr 6. PMID 23570660
- [Background] Doi K, Tanaka S, Iida H, Eto H, Kato H, Aoi N, Kuno S, Hirohi T, Yoshimura K. Stromal vascular fraction isolated from lipo-aspirates using an automated processing system: bench and bed analysis. J Tissue Eng Regen Med. 2013 Nov;7(11):864-70. doi: 10.1002/term.1478. Epub 2012 Mar 22. PMID 22438241
- [Background] Williams SK, Kosnik PE, Kleinert LB, Vossman EM, Lye KD, Shine MH. Adipose stromal vascular fraction cells isolated using an automated point of care system improve the patency of expanded polytetrafluoroethylene vascular grafts. Tissue Eng Part A. 2013 Jun;19(11-12):1295-302. doi: 10.1089/ten.TEA.2012.0318. Epub 2013 Mar 15. PMID 23350681
- [Background] Hernigou P, Flouzat Lachaniette CH, Delambre J, Zilber S, Duffiet P, Chevallier N, Rouard H. Biologic augmentation of rotator cuff repair with mesenchymal stem cells during arthroscopy improves healing and prevents further tears: a case-controlled study. Int Orthop. 2014 Sep;38(9):1811-8. doi: 10.1007/s00264-014-2391-1. Epub 2014 Jun 7. PMID 24913770